CLINICAL TRIAL: NCT05783297
Title: Midwest TXTXT Scale up of an Evidence-Based Intervention to Promote HIV Medication Adherence
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: University of Illinois at Chicago (Other); KC Care Health Center (Other); Eskenazi Health (Other); Corktown Health Center (Unknown); Howard Brown Health Center (Other); University of Cincinnati (Other); Indiana University (Other); Duke University (Other); Amity Medical Group (Unknown); Valley AIDS Council (Other); Baylor College of Medicine (Other); AIDS Healthcare Foundation (Other); Comprehensive Care Center of Southwest Louisiana (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: U01PS005214 (NIH)
Record Dates: First submitted 2023-01-17; First posted 2023-03-24 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The proposed research uses a cluster randomized controlled trial design to evaluate the effectiveness of TXTXT intervention on adherence and viral load suppression at 3- and 6- months post intervention initiation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparison (Active Comparator): Clinics randomized to the comparison arm will have participants receive standard of care ART adherence support for 3 months, and will receive the TXTXT intervention for 3 months. The standard of care for ART adherence across clinic sites consists of routine follow-up from assigned case managers for appointment reminders and adherence counseling at scheduled visits .
  Interventions: Behavioral: Standard of Care
- Intervention (Experimental): Clinics randomized to the intervention arm will have participants complete a 6-month intervention period. Clinics will sign up eligible participants to receive automated SMS messages from the Dimagi CommCare platform during the participant's baseline study visit. Participants will have the option to tailor the message content based on their own preferences and will be able to select to receive messages in English or in Spanish, the time the messages are delivered, and frequency of messages. Clinic staff will enter this information in the Dimagi CommCare platform, and then test receipt of text messages by the participant before they complete this baseline visit.
  Interventions: Behavioral: Treatment Text (TXTXT)

INTERVENTIONS:
Behavioral: Treatment Text (TXTXT) — This study will test a tailored, personalized SMS text message reminder intervention to improve adherence to ART among non-adherent youth and young adults with HIV. Participants will use their own cell phones for receipt of the intervention. Participants will have the option to choose a tailored personalized message that may be changed as requested throughout the 6-month intervention period. Participants will be asked to send a text message response indicating that that have successfully (or not) taken their meds per schedule. No identifying patient information will be included in the SMS text to protect patient confidentiality.
  Arms: Intervention
Behavioral: Standard of Care — Standard of care ART adherence support includes adherence counseling during visits scheduled at least twice annually and appointment reminders.
  Arms: Comparison

SUMMARY:
This research study uses a cluster randomized controlled trial design to evaluate the effectiveness of Treatment Text (TXTXT) intervention on adherence and viral load suppression at 3- and 6- months post intervention initiation for youth and young adults with HIV. A total of 12 clinics will be randomized into one of the following two conditions:

1. Comparison Arm (n=6 clinics)- Clinics randomized to the comparison arm will have participants receive the standard of care for 3 months, followed by a 3-month intervention period.
2. Intervention Arm (n=6 clinics)- Clinics randomized to the intervention arm will have participants receive the TXTXT intervention for 6 months.

DETAILED DESCRIPTION:
In this study investigators propose to use implementation science (IS) to scale up and evaluate the TXTXT evidence-based intervention (EBI) as an effective strategy to increase ART adherence and retention in HIV care, ultimately leading to a suppression of viral load in youth and young adults with HIV (YYALH) participating in the intervention. Investigators hypothesize that participants who complete the TXTXT intervention will demonstrate a clinically meaningful increase in ART adherence, viral suppression, and sustained retention in care. Additionally, investigators hypothesize that the implementation of TXTXT will reach ≥80% of the intended participants, will be fully adopted by ≥80% of clinic partners, and will achieve ≥90% ratings of satisfaction and acceptability. Investigators will use mixed methods to complete the study aims: 1) determine the real-world efficacy of a regional scale up of an EBI - TXTXT - among poorly adherent YYALH, aged 16-35 years, on our primary outcomes: adherence and viral load suppression at 3-month post initiation of the intervention; and secondary outcome: retention in HIV care at 6- and 12-months post baseline, and 2) apply the Consolidated Framework for Implementation Research (CFIR) to describe the implementation process and identify barriers and facilitators needed to be addressed; and measure implementation outcomes of the TXTXT intervention using the RE-AIM framework (Reach, Efficacy, Adoption, Implementation, Maintenance). Investigators will conduct a cluster randomized controlled trial to evaluate the intervention effectiveness (i.e., ART adherence, viral load suppression) at 3- and 6-months post-initiation of the intervention. Twelve clinic sites with the ability to enroll up to 50 participants at each site (N=600 participants total) will be trained to administer the TXTXT intervention. Sites will be randomized to either start the intervention immediately (i.e., intervention arm) or waitlisted to start at 3 months post baseline (i.e., comparison arm). In the comparison arm, the study will compare pre-post differences in adherence at 3- and 6-months post baseline. Last, investigators will evaluate retention in HIV care, viral suppression, and sustained impact of the intervention at 6 months and 12 months post baseline for all study participants.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with HIV-infection and on ART regimen for at least one month
2. Between 16-35 years of age
3. Have a viral load ≥200c/mL and/or report poor adherence (<90% of pills taken in the last 30 days)
4. Able to receive text messages
5. Can provide informed consent for research component
6. Current patient patient of a participating clinic

Exclusion Criteria:

1. Participant is unable to give informed consent
2. Participant is participating in another study related to ART adherence

Participants outside of the age range (16-35) will be excluded from the study because this study specifically focuses on youth and young adults living with HIV as they are more likely to disengage from care, delay initiation of ART, and have lower rates of virologic suppression compared to adult populations.

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
HIV-1 RNA Viral Load | Up to 12 months
  A documented viral load measured by nucleic acid test (NAT) less than (<) 200 copies/mL will be considered virally suppressed. The minimum value is 20 copies/mL and the maximum is 10,000,000 copies/mL. A higher value indicates a worse outcome. Time frame: 6 months, 12 months.
HIV Medication Adherence | Up to 12 months
  Medication adherence will be measured via self-reported visual analog scale. The minimum value is 0% and the maximum value is 100%. A higher value indicates a better outcome. Adherence will be considered reporting greater than or equal to 90% on self-reported visual analog scale and non- adherence categorized at less than 90%. Time frame: 3 months, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Amy Johnson, PhD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (12):
- United States (12):
  - AIDS Healthcare Foundation, Fort Lauderdale, Florida
  - University of Illinois at Chicago, Chicago, Illinois
  - Howard Brown Health, Chicago, Illinois
  - Eskenazi Health, Indianapolis, Indiana
  - Indiana University, Indianapolis, Indiana
  - Comprehensive Care Center of Southwest Louisiana, Lake Charles, Louisiana
  - Corktown Health Center, Detroit, Michigan
  - KC Care Health Center, Kansas City, Missouri
  - Duke University, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Baylor College of Medicine, Houston, Texas
  - Valley AIDS Council, McAllen, Texas

IPD SHARING:
Plan to Share IPD: Yes
We will share restricted de-identified datasets with those who initiate a data request and data sharing agreement via the PI (Dr. Amy Johnson).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will be available by request within 6-months of the trial end date.
Access Criteria: Completion of a data request form and execution of a data sharing form with the study PI and PI's institution.

REFERENCES:
- [Background] Centers for Disease Control and Prevention. Diagnoses of HIV infection in the United States and dependent areas, 2019. (2019).
- [Background] Denning, P. & DiNenno, E. in XVIII international AIDS conference.
- [Background] Maulsby C, Millett G, Lindsey K, Kelley R, Johnson K, Montoya D, Holtgrave D. HIV among Black men who have sex with men (MSM) in the United States: a review of the literature. AIDS Behav. 2014 Jan;18(1):10-25. doi: 10.1007/s10461-013-0476-2. PMID 23620241
- [Background] Bangsberg DR. Less than 95% adherence to nonnucleoside reverse-transcriptase inhibitor therapy can lead to viral suppression. Clin Infect Dis. 2006 Oct 1;43(7):939-41. doi: 10.1086/507526. Epub 2006 Aug 23. PMID 16941380
- [Background] Cohen MS, Chen YQ, McCauley M, Gamble T, Hosseinipour MC, Kumarasamy N, Hakim JG, Kumwenda J, Grinsztejn B, Pilotto JH, Godbole SV, Mehendale S, Chariyalertsak S, Santos BR, Mayer KH, Hoffman IF, Eshleman SH, Piwowar-Manning E, Wang L, Makhema J, Mills LA, de Bruyn G, Sanne I, Eron J, Gallant J, Havlir D, Swindells S, Ribaudo H, Elharrar V, Burns D, Taha TE, Nielsen-Saines K, Celentano D, Essex M, Fleming TR; HPTN 052 Study Team. Prevention of HIV-1 infection with early antiretroviral therapy. N Engl J Med. 2011 Aug 11;365(6):493-505. doi: 10.1056/NEJMoa1105243. Epub 2011 Jul 18. PMID 21767103
- [Background] Gardner EM, McLees MP, Steiner JF, Del Rio C, Burman WJ. The spectrum of engagement in HIV care and its relevance to test-and-treat strategies for prevention of HIV infection. Clin Infect Dis. 2011 Mar 15;52(6):793-800. doi: 10.1093/cid/ciq243. PMID 21367734
- [Background] Reisner SL, Mimiaga MJ, Skeer M, Perkovich B, Johnson CV, Safren SA. A review of HIV antiretroviral adherence and intervention studies among HIV-infected youth. Top HIV Med. 2009 Feb-Mar;17(1):14-25. PMID 19270345
- [Background] Agwu AL, Fleishman JA, Korthuis PT, Siberry GK, Ellen JM, Gaur AH, Rutstein R, Gebo KA; HIV Research Network. Disparities in antiretroviral treatment: a comparison of behaviorally HIV-infected youth and adults in the HIV Research Network. J Acquir Immune Defic Syndr. 2011 Sep 1;58(1):100-7. doi: 10.1097/QAI.0b013e31822327df. PMID 21637114
- [Background] Giordano TP, Visnegarwala F, White AC Jr, Troisi CL, Frankowski RF, Hartman CM, Grimes RM. Patients referred to an urban HIV clinic frequently fail to establish care: factors predicting failure. AIDS Care. 2005 Aug;17(6):773-83. doi: 10.1080/09540120412331336652. PMID 16036264
- [Background] Lee L, Yehia BR, Gaur AH, Rutstein R, Gebo K, Keruly JC, Moore RD, Nijhawan AE, Agwu AL; HIV Research Network. The Impact of Youth-Friendly Structures of Care on Retention Among HIV-Infected Youth. AIDS Patient Care STDS. 2016 Apr;30(4):170-7. doi: 10.1089/apc.2015.0263. Epub 2016 Mar 16. PMID 26983056
- [Background] Minniear TD, Gaur AH, Thridandapani A, Sinnock C, Tolley EA, Flynn PM. Delayed entry into and failure to remain in HIV care among HIV-infected adolescents. AIDS Res Hum Retroviruses. 2013 Jan;29(1):99-104. doi: 10.1089/AID.2012.0267. Epub 2012 Nov 7. PMID 23033848
- [Background] Ryscavage P, Anderson EJ, Sutton SH, Reddy S, Taiwo B. Clinical outcomes of adolescents and young adults in adult HIV care. J Acquir Immune Defic Syndr. 2011 Oct 1;58(2):193-7. doi: 10.1097/QAI.0b013e31822d7564. PMID 21826014
- [Background] Torian LV, Wiewel EW. Continuity of HIV-related medical care, New York City, 2005-2009: Do patients who initiate care stay in care? AIDS Patient Care STDS. 2011 Feb;25(2):79-88. doi: 10.1089/apc.2010.0151. PMID 21284498
- [Background] Vijayan T, Benin AL, Wagner K, Romano S, Andiman WA. We never thought this would happen: transitioning care of adolescents with perinatally acquired HIV infection from pediatrics to internal medicine. AIDS Care. 2009 Oct;21(10):1222-9. doi: 10.1080/09540120902730054. PMID 20024697
- [Background] Yehia BR, Fleishman JA, Metlay JP, Moore RD, Gebo KA. Sustained viral suppression in HIV-infected patients receiving antiretroviral therapy. JAMA. 2012 Jul 25;308(4):339-42. doi: 10.1001/jama.2012.5927. No abstract available. PMID 22820781
- [Background] Zanoni BC, Mayer KH. The adolescent and young adult HIV cascade of care in the United States: exaggerated health disparities. AIDS Patient Care STDS. 2014 Mar;28(3):128-35. doi: 10.1089/apc.2013.0345. PMID 24601734
- [Background] MacDonell K, Naar-King S, Huszti H, Belzer M. Barriers to medication adherence in behaviorally and perinatally infected youth living with HIV. AIDS Behav. 2013 Jan;17(1):86-93. doi: 10.1007/s10461-012-0364-1. PMID 23142855
- [Background] Garofalo R, Kuhns LM, Hotton A, Johnson A, Muldoon A, Rice D. A Randomized Controlled Trial of Personalized Text Message Reminders to Promote Medication Adherence Among HIV-Positive Adolescents and Young Adults. AIDS Behav. 2016 May;20(5):1049-59. doi: 10.1007/s10461-015-1192-x. PMID 26362167
- [Background] Project, H. A. P. R. S. (ed Centers for Disease Control and Prevention) https://www.cdc.gov/hiv/research/interventionresearch/compendium/index.html (2020).
- [Background] Fauci AS, Redfield RR, Sigounas G, Weahkee MD, Giroir BP. Ending the HIV Epidemic: A Plan for the United States. JAMA. 2019 Mar 5;321(9):844-845. doi: 10.1001/jama.2019.1343. No abstract available. PMID 30730529
- [Background] Hosek SG, Harper GW, Domanico R. Predictors of medication adherence among HIV-infected youth. Psychol Health Med. 2005 May;10(2):166-179. doi: 10.1080/1354350042000326584. PMID 25705113
- [Background] Centers for Disease Control and Prevention. Vol. 29 (ed Department of Health and Human Services) (Division of HIV/AIDS Prevention, National Center for HIV/AIDS, Viral Hepatitis, STD, and TB Prevention, Centers for Disease Control and Prevention (CDC), U.S. Department of Health and Human Services, Atlanta, GA, 2018).
- [Background] Collins CB Jr, Sapiano TN. Lessons Learned From Dissemination of Evidence-Based Interventions for HIV Prevention. Am J Prev Med. 2016 Oct;51(4 Suppl 2):S140-7. doi: 10.1016/j.amepre.2016.05.017. Epub 2016 Jul 9. PMID 27402185
- [Background] Bauermeister JA, Tross S, Ehrhardt AA. A review of HIV/AIDS system-level interventions. AIDS Behav. 2009 Jun;13(3):430-48. doi: 10.1007/s10461-008-9379-z. Epub 2008 Mar 28. PMID 18369722
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Lambdin BH, Cheng B, Peter T, Mbwambo J, Apollo T, Dunbar M, Udoh IC, Cattamanchi A, Geng EH, Volberding P. Implementing Implementation Science: An Approach for HIV Prevention, Care and Treatment Programs. Curr HIV Res. 2015;13(3):244-9. doi: 10.2174/1570162x1303150506185423. PMID 25986374
- [Background] Whiteley LB, Olsen EM, Haubrick KK, Odoom E, Tarantino N, Brown LK. A Review of Interventions to Enhance HIV Medication Adherence. Curr HIV/AIDS Rep. 2021 Oct;18(5):443-457. doi: 10.1007/s11904-021-00568-9. Epub 2021 Jun 21. PMID 34152554
- [Background] Zullig LL, Deschodt M, Liska J, Bosworth HB, De Geest S. Moving from the Trial to the Real World: Improving Medication Adherence Using Insights of Implementation Science. Annu Rev Pharmacol Toxicol. 2019 Jan 6;59:423-445. doi: 10.1146/annurev-pharmtox-010818-021348. Epub 2018 Aug 20. PMID 30125127
- [Background] Glasgow RE, Emmons KM. How can we increase translation of research into practice? Types of evidence needed. Annu Rev Public Health. 2007;28:413-33. doi: 10.1146/annurev.publhealth.28.021406.144145. PMID 17150029
- [Background] Bandura A. Social cognitive theory: an agentic perspective. Annu Rev Psychol. 2001;52:1-26. doi: 10.1146/annurev.psych.52.1.1. PMID 11148297
- [Background] Hedeker, D. in Encyclopedia of Statistics in Behavioral Science (eds B. Everitt & D. Howell) (Wiley, 2005).
- [Background] Diggle, P., Liang, K.-Y. & Zeger, S. L. Longitudinal data analysis. New York: Oxford University Press 5, 13 (1994).
- [Background] Lewis MA, Harshbarger C, Bann C, Burrus O, Peinado S, Garner BR, Khavjou O, Shrestha RK, Karns S, Borkowf CB, Zulkiewicz BA, Ortiz A, Galindo CA, DallaPiazza M, Holm P, Marconi VC, Somboonwit C, Swaminathan S; Positive Health Check Study Team. Positive Health Check evaluation: A type 1 hybrid design randomized trial to decrease HIV viral loads in patients seen in HIV primary care. Contemp Clin Trials. 2020 Sep;96:106097. doi: 10.1016/j.cct.2020.106097. Epub 2020 Jul 29. PMID 32738408
- [Background] Mugavero MJ, Westfall AO, Zinski A, Davila J, Drainoni ML, Gardner LI, Keruly JC, Malitz F, Marks G, Metsch L, Wilson TE, Giordano TP; Retention in Care (RIC) Study Group. Measuring retention in HIV care: the elusive gold standard. J Acquir Immune Defic Syndr. 2012 Dec 15;61(5):574-80. doi: 10.1097/QAI.0b013e318273762f. PMID 23011397
- [Background] Health Resources & Services Administration. HIV/AIDS Bureau Performance Measures. (2019).
- [Background] Ahn, C., Heo, M. & Zhang, S. Sample Size Calculations for Clustered and Longitudinal Outcomes in Clinical Research. 1 edn, 223-225 (Chapman and Hall, 2015).
- [Background] Keith RE, Crosson JC, O'Malley AS, Cromp D, Taylor EF. Using the Consolidated Framework for Implementation Research (CFIR) to produce actionable findings: a rapid-cycle evaluation approach to improving implementation. Implement Sci. 2017 Feb 10;12(1):15. doi: 10.1186/s13012-017-0550-7. PMID 28187747
- [Background] SocioCultural Research Consultants, L. (Los Angeles, CA, 2018)
- [Background] Hsieh HF, Shannon SE. Three approaches to qualitative content analysis. Qual Health Res. 2005 Nov;15(9):1277-88. doi: 10.1177/1049732305276687. PMID 16204405
- [Background] Tinsley, H. E. & Weiss, D. J. in Handbook of applied multivariate statistics and mathematical modeling 95-124 (Elsevier, 2000).
- [Background] Breimaier HE, Heckemann B, Halfens RJ, Lohrmann C. The Consolidated Framework for Implementation Research (CFIR): a useful theoretical framework for guiding and evaluating a guideline implementation process in a hospital-based nursing practice. BMC Nurs. 2015 Aug 12;14:43. doi: 10.1186/s12912-015-0088-4. eCollection 2015. PMID 26269693

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT05783297/Prot_SAP_ICF_000.pdf